CLINICAL TRIAL: NCT04861025
Title: Perception of Users and Healthcare Professionals on Siderails Prescription as a Measure of Physical Restraint
Brief Title: Siderails as a Measure of Physical Restraint. GERBAR Trial
Acronym: GERBAR
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-19
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-03

CONDITIONS: Restraint, Physical; Aged; Aged, 80 and Over; Patient Safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Users Group: Patients admitted to any Hospitalization Unit belonging to Geriatrics Department
- Health Professionals Group: All health professionals working at some Hospitalization Unit belonging to CSAPG Institution

SUMMARY:
There is a controversy about if siderails should be considered as a method of physical restraint in older hospitalized patients. This study aims to investigate the opinion of older patients and health professionals about this controversy.

DETAILED DESCRIPTION:
Aim: to know the perception of older patients and health professionals regarding bedrails using as a method of physical restraint.

Design: quasi-experimental study ("before-after").

Duration: 13 months

Sample:

Two samples will be recruited: one from older patients who are hospitalized at Geriatric Hospitalization Units participating in the study, and the other one including all health professionals working at the 3 hospitals which belong to the Consorci Sanitari de l'Alt Penedès i Garraf.

Sample size:

Being the main objective of the study the estimation of a proportion (proportion of users who consider the siderails as a method of physical restraint), and having a preliminary estimation (65%) of this perception in older patients from a preliminary study, we calculated a sample size of 270 participants, considering a confidence level of 95% with a precision +/- 6%, and a necessary replacement rate of 10%. In the case of healthcare professionals, we calculated a sample size of 85 participants, considering an estimated proportion of 30%, a confidence level of 95% with a precision of +/- 10%, and a necessary replacement proportion of 5%.

Procedures:

In the sample of health professionals, a single online survey questionnaire is expected in month 1 with the purpose of knowing the health professional's perception of siderails as a method of physical restraint.

Once the health professionals' evaluations are finalized, the older patient recruitment will start. A baseline evaluation (interview) will be performed within days 0-2 of admission at the hospitalization unit. In this evaluation, basal data, the perception of bedrails as a method of physical restraint, and a register of patient's desire on using bedrails during their hospitalization will be collected. Then, two follow-up evaluations (days +1 and +2 from baseline evaluation) will be done to record the use of the siderails.

Participants' recruitment:

After the first register of use of bedrails at the Geriatric Hospitalization Units, the researchers will inform the health professionals about the objectives and design of the study, and compliance with the inclusion and exclusion criteria will be verified. If the health professional agrees to participate, the information sheet will be delivered and the informed consent will be collected. All health professionals will complete the survey questionnaire individually, anonymously, and in electronic format.

Older patient's recruitment and their baseline assessment will take place on the same day. The collaborating investigator of the study will invite all those users who undergo the clinical admission interview in the participating hospitalization unit to participate in the study, and within the first two days of admission. Once the study admission criteria have been confirmed, and the participant's informed consent has been obtained, the baseline interview will be carried out. In this interview, the user's perception of the bedrails and their willingness to use them during their hospitalization will be registered. Subsequently, the collaborator will communicate the patient's desire to the nursing team orally and registering the desire at the clinical record.

In the case of participants with Pfeiffer test ≥ 5 errors or a positive result for the Confusional Assessment Method test, a patient's relative or accompanying person will also be interviewed. In the event that the participant is not clinically stable to be interviewed according to the criteria of the interviewer, the interview will be carried out exclusively with the family member or accompanying person.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1 (Healthcare professionals):

   a. Any health professional (nursing assistant, nurse, doctor...) who belons to CSAPG Institution.
2. Group 2 (Users):

   1. Patient aged 65 or more years admitted to one of the participating Hospitalization Units belonging to Geriatrics Department.

Exclusion Criteria:

1. Group 1 (Healthcare professionals):

   a. Refusal to participate in the study.
2. Group 2 (Users):

   1. Users in palliative sedation or with short /very short life expectancy.
   2. Inability to consent and absence of a legal representative.
   3. Refusal to participate in the study.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All older patients admitted to Hospitalization Units belonging to Geriatrics Department.
  All health professionals working at a Secondary Care Center.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients considering siderails as a physical restraint method | Baseline
  Proportion of older patients (regard to all of hospitalized older patients) who consider siderails as a physical restraint's method
Proportion of health professionals considering siderails as a physical restraint method | Baseline
  Proportion of health professionals (regard to all health professionals working at the hospital) who consider siderails as a physical restraint's method

SECONDARY OUTCOMES:
Factors associated to prescription of siderails by health professionals | Hospital discharge (assessed up to day 180)
  Factors associated to prescription of siderails by health professionals
Factors associated to prescription of siderails by hospitalized patients | Hospital discharge (assessed up to day 180)
  Factors associated to prescription of siderails by hospitalized patients

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Macho Perez, MD, Principal Investigator — Consorci Sanitari d'Alt Penedès i Garraf
Locations (1):
- Consorci Sanitari d'Alt Penedès i Garraf, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research proposels and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.

REFERENCES:
- [Background] Macho-Perez O, Arroyo-Huidobro M, Gimenez Buendia MDC, Galvez-Barron C. [Does the healthcare user consider rails as physical subjugation?]. Rev Esp Geriatr Gerontol. 2021 Jan-Feb;56(1):59-60. doi: 10.1016/j.regg.2020.06.008. Epub 2020 Oct 17. No abstract available. Spanish. PMID 33081978
- [Result] Galvez-Barron C, Gonzalez-De Luna A, Perez-Lopez C, Macho-Perez O. Cross-sectional survey of healthcare professionals' perceptions of bedrails as a measure of physical restraint in the hospital setting. Age Ageing. 2025 Jan 6;54(1):afaf002. doi: 10.1093/ageing/afaf002. PMID 39851241